CLINICAL TRIAL: NCT00335738
Title: A Study of Unilateral Retinoblastoma With and Without Histopathologic High-Risk Features and the Role of Adjuvant Chemotherapy
Brief Title: Vincristine, Carboplatin, and Etoposide or Observation Only in Treating Patients Who Have Undergone Surgery for Newly Diagnosed Retinoblastoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARET0332; NCI-2009-00423 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000483043 (Other: Clinical Trials.gov); U10CA098543 (NIH); COG-ARET0332 (Other: Children's Oncology Group)
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2018-03

CONDITIONS: Intraocular Retinoblastoma
MeSH Terms: interventions — Vincristine; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (identified by central review as high risk) (Experimental): Includes patients who may or may not require chemotherapy. Patients who require chemotherapy receive vincristine IV and carboplatin IV over 1 hour on day 1 and etoposide IV over 1 hour on days 1 and 2. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity and patients who complete chemotherapy are followed after completion of therapy periodically for at least 5 years. Patients who do not require chemotherapy undergo observation periodically for at least 5 years.
  Interventions: Drug: liposomal vincristine sulfate; Drug: carboplatin; Drug: etoposide
- Group 2 (identified by central review as not high risk) (No Intervention): Patients undergo observation periodically for at least 5 years.

INTERVENTIONS:
Drug: liposomal vincristine sulfate — Given IV
  Other Names: liposomal vincristine; Marqibo; vincristine liposomal; vincristine sulfate liposome injection
  Arms: Group 1 (identified by central review as high risk)
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
  Arms: Group 1 (identified by central review as high risk)
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
  Arms: Group 1 (identified by central review as high risk)

SUMMARY:
This phase III trial is studying vincristine, carboplatin, and etoposide to see how well they work compared to observation only in treating patients who have undergone surgery for newly diagnosed retinoblastoma. Drugs used in chemotherapy, such as vincristine, carboplatin, and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) after surgery may kill any tumor cells that remain after surgery. Sometimes, after surgery, no additional treatment is needed for the tumor until it progresses. In this case, observation may be sufficient.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Prospectively determine the prevalence of high-risk histopathologic features, such as choroidal involvement, optic nerve invasion, and scleral and anterior segment involvement, in patients with newly diagnosed unilateral retinoblastoma who have undergone enucleation.

II. Demonstrate that patients without certain high-risk features can be successfully treated with enucleation alone by estimating the event-free survival (EFS) (where an event is defined as the occurrence of extraocular or metastatic disease) and overall survival (OS).

III. Estimate the EFS and OS of patients with specific high-risk features who are uniformly treated with adjuvant chemotherapy comprising vincristine, carboplatin, and etoposide.

IV. Estimate the incidence of toxicities associated with the proposed adjuvant chemotherapy regimen.

OUTLINE: This is a prospective, nonrandomized, multicenter study. Patients are assigned to 1 of 2 groups according to presence of high-risk histopathologic features.

GROUP 1 (high-risk features): Patients receive vincristine IV and carboplatin IV over 1 hour on day 1 and etoposide IV over 1 hour on days 1 and 2. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

GROUP 2 (no high-risk features): Patients undergo observation periodically for at least 5 years.

GROUP 3 (no consensus regarding high risk features can be reached): Patients undergo Group 1 chemotherapy or observation according to institutional high-risk feature assessment.

After completion of study treatment, patients in group 1 are followed periodically for at least 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed unilateral retinoblastoma
* Underwent enucleation as primary therapy within the past 5 weeks

  * Must enroll and submit pathology slides within 21 days of enucleation
  * Adjuvant chemotherapy must begin within 35 days after enucleation
* Disease with or without high-risk histopathologic features

  * High-risk features are defined as any of the following:

    * Posterior uveal invasion (includes choroidal invasion)
    * Any degree of concomitant choroid and/or optic nerve involvement
    * Tumor involving the optic nerve posterior to the lamina cribrosa as an independent finding
    * Scleral invasion
    * Anterior chamber seeding
    * Ciliary body infiltration
    * Iris infiltration
* No evidence of extraocular retinoblastoma clinically, by CT scan, or by MRI of the brain and orbits with and without gadolinium
* No tumor at the cut end of the optic nerve on any eye enucleated as evidenced by histologic examination prior to study entry
* No systemic metastases as evidenced by bone marrow scan, bone scan, or any other additional test at study entry
* Lansky performance status 50-100%
* Hemoglobin > 8 g/dL
* Absolute neutrophil count ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine adjusted according to age as follows:

  * No greater than 0.4 mg/dL (≤ 5 months)
  * No greater than 0.5 mg/dL (6 months -11 months)
  * No greater than 0.6 mg/dL (1 year-23 months)
  * No greater than 0.8 mg/dL (2 years-5 years)
  * No greater than 1.0 mg/dL (6 years-9 years)
  * No greater than 1.2 mg/dL (10 years-12 years)
  * No greater than 1.4 mg/dL (13 years and over [female])
  * No greater than 1.5 mg/dL (13 years to 15 years [male])
  * No greater than 1.7 mg/dL (16 years and over [male])
* Creatinine clearance or radioisotope glomerular filtration rate at least 70 mL/min
* Bilirubin ≤ 1.5 times upper limit of normal (ULN) for age
* AST or ALT < 2.5 times ULN for age
* No prior therapy other than enucleation
* No prior chemotherapy

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 331 (Actual)
Dates: Start 2005-12; Primary Completion 2011-09 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murali Chintagumpala, MD, Principal Investigator — Children's Oncology Group
Locations (56):
- United States (48):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - Children's Oncology Group, Arcadia, California
  - Southern California Permanente Medical Group, Downey, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - University of California San Francisco Medical Center-Parnassus, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lombardi Comprehensive Cancer Center at Georgetown University, Washington D.C., District of Columbia
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - University of Illinois, Chicago, Illinois
  - Childrens Memorial Hospital, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Maine Children's Cancer Program, Scarborough, Maine
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Brooklyn Hospital Center, Brooklyn, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Medical Center of Dayton, Dayton, Ohio
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Childrens Hospital-King's Daughters, Norfolk, Virginia
  - Marshfield Clinic, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (3):
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (2):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Hospital Sainte-Justine, Montreal, Quebec
- L V Prasad Eye Institute, Hyderabad, India
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch

REFERENCES:
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 (Identified by Central Review as High Risk) | Group 2 (Identified by Central Review as Not High Risk)
Started | 108 | 223
Completed | 97 | 219
Not Completed | 11 | 4
Not completed — Physician Decision | 6 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Ineligible | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Group 1 (High Risk): Patients receive liposomal vincristine sulfate IV aged based dosage (Pts < 36 mos: 0.05 mg/kg, Pts > 36 mos: 1.5 mg/m2, max dose 2 MG) given IV or infusion on day 1, carboplatin aged based dosage (Pts < 36 mos: 18.6 mg/kg Pts > 36 mos: 560 mg/m2) IV on day 1, and Etoposide aged based dosage (Pts < 36 mos: 5 mg/kg, Pts > 36 mos: 150 mg/m2) IV on days 1 and 2. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  liposomal vincristine sulfate: Given IV
  carboplatin: Given IV
  etoposide: Given IV
- Group 2 (Not High Risk): Patients undergo observation periodically for at least 5 years.
- Total: Total of all reporting groups
Arm/Group | Group 1 (High Risk) | Group 2 (Not High Risk) | Total
Number analyzed (Participants) | 108 | 223 | 331
Age, Continuous [Median (Full Range); unit: years] | 2 [0 to 6] | 1 [0 to 6] | 2 [0 to 6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 107 | 159
  Male | 56 | 116 | 172
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 32 | 56
  Not Hispanic or Latino | 82 | 181 | 263
  Unknown or Not Reported | 2 | 10 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 37 | 63 | 100
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 8 | 17 | 25
  White | 43 | 108 | 151
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 18 | 34 | 52
Region of Enrollment [Number; unit: participants]
  United States | 65 | 144 | 209
  New Zealand | 1 | 7 | 8
  India | 32 | 55 | 87
  Mexico | 1 | 0 | 1
  Canada | 3 | 7 | 10
  Australia | 6 | 8 | 14
  Bangladesh | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS)
Description: EFS distributions will be estimated by the Kaplan-Meier method for patients with high risk features according to central review and treated with adjuvant chemotherapy and separately for subjects with central review recommendation of enucleation alone.
Time Frame: At 2 years
Population: Only eligible patients are considered in the characterization of EFS at 2 years.
Measure: Number (95% Confidence Interval); unit: Estimated Probability
Arm/Group | Group 1 (Identified by Central Review as High Risk) | Group 2 (Identified by Central Review as Not High Risk)
Number analyzed (Participants) | 89 | 235
Estimated Probability | 0.9394 [0.8606 to 0.9743] | 0.9953 [0.9671 to 0.9993]

2. Primary Outcome: Overall Survival (OS)
Description: OS distributions will be estimated by the Kaplan-Meier method for patients with high risk features according to central review and treated with adjuvant chemotherapy and separately for subjects with central review recommendation of enucleation alone.
Time Frame: At 2 Years
Population: Only eligible patients are considered for this outcome measure. This is calculated as the total number of patients enrolled in each group with the number ineligible in each group subtracted as reported on the participant flow template.
Measure: Number (95% Confidence Interval); unit: Estimated Probability
Arm/Group | Group 1 (Identified by Central Review as High Risk) | Group 2 (Identified by Central Review as Not High Risk)
Number analyzed (Participants) | 89 | 235
Estimated Probability | 0.9628 [0.8890 to 0.9878] | 1 [1 to 1]

3. Secondary Outcome: Toxicity As Assessed By the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: Number of patients assigned chemotherapy who experienced grade 3 or higher CTC AE toxicity.
Time Frame: During planned six cycles of chemotherapy
Population: Adverse experiences as coded using CTC AE version 4 were collected only for patients who received chemotherapy according to protocol guidelines. Of the 105 eligible patients with high risk features, ninety-three (93) were given protocol chemotherapy based on the assessment of the central pathology review, as described in section 4 of the ARET0332.
Measure: Number; unit: participants
Arm/Group | Group 1 (Identified by Central Review as High Risk)
Number analyzed (Participants) | 93
participants | 19

4. Secondary Outcome: Pathological Features Present At Diagnosis - Posterior Uveal Invasion (PVI)
Description: Proportion of patients who had posterior uveal invasion at enrollment.
Time Frame: At enrollment
Population: Central review of the biological materials for this aim was available on only 313 patients. This outcome measure is calculated by combing all groups as characterized in the Patient Flow.
Measure: Number (95% Confidence Interval); unit: Proportion of patients with PVI
Groups:
- All Patients: This outcome measure is calculated by combining all groups as defined in the trials record.
Arm/Group | All Patients
Number analyzed (Participants) | 313
Proportion of patients with PVI | 0.24 [0.19 to 0.29]

5. Secondary Outcome: Pathological Features Present At Diagnosis - Tumor Involving the Optic Nerve Posterior to the Lamina Cribrosa (LC) as an Independent Finding
Description: Proportion of patients with tumor involving the optic nerve posterior to the lamina cribrosa as an independent.
Time Frame: At enrollment
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Proportion of patients with LC
Arm/Group | All Patients
Number analyzed (Participants) | 313
Proportion of patients with LC | 0.16 [0.12 to 0.21]

6. Secondary Outcome: Pathological Features Present at Diagnosis - Scleral Invasion (SI)
Description: Proportion of patients that had scleral invasion at enrollment.
Time Frame: At enrollment
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Proportion of patients with SI
Arm/Group | All Patients
Number analyzed (Participants) | 313
Proportion of patients with SI | 0.016 [0.0052 to 0.037]

7. Secondary Outcome: Pathological Features Present At Diagnosis - Anterior Chamber Seeding (ACS)
Description: Proportion of patients who had anterior chamber seeding at enrollment.
Time Frame: At enrollment
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Proportion of patients with ACS
Arm/Group | All Patients
Number analyzed (Participants) | 313
Proportion of patients with ACS | 0.045 [0.025 to 0.074]

8. Secondary Outcome: Pathological Features Present At Diagnosis - Iris Infiltration (II)
Description: Proportion of patients who had iris infiltration at enrollment.
Time Frame: At enrollment
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Proportion of patients with II
Arm/Group | All Patients
Number analyzed (Participants) | 313
Proportion of patients with II | 0.029 [0.013 to 0.054]

9. Secondary Outcome: Pathological Features Present At Diagnosis - Ciliary Body Infiltration (CBI)
Description: Proportion of patients who had ciliary body infiltration at enrollment.
Time Frame: At Enrollment
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Proportion of patients with CBI
Arm/Group | All Patients
Number analyzed (Participants) | 313
Proportion of patients with CBI | 0.019 [0.0071 to 0.041]

ADVERSE EVENTS:
Description: Adverse experiences as coded using CTC AE version 4 were collected only for patients who received chemotherapy according to protocol guidelines. Of the 105 eligible patients with high risk features, ninety-three (93) were given protocol chemotherapy based on the assessment of the central pathology review, as described in section 4 of the ARET0332 protocol.
Arm/Group | Group 1 (Identified by Central Review as High Risk) | Group 2 (Identified by Central Review as Not High Risk)
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/0
Other Adverse Events (participants affected / at risk) | 19/93 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Identified by Central Review as High Risk) (N=93) | Group 2 (Identified by Central Review as Not High Risk) (N=0)
Alanine aminotransferase increased (Investigations) | 1 | 0
Anaphylaxis (Immune system disorders) | 5 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 9 | 0
Headache (Nervous system disorders) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 2 | 0
Neutrophil count decreased (Investigations) | 6 | 0
Otitis media (Infections and infestations) | 1 | 0
Platelet count decreased (Investigations) | 4 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0

LIMITATIONS AND CAVEATS:
The COG SDC reviewed the NLM notification related to ct.gov AE/SAE reporting. The information in 'Additional Description' is accurate with respect to data supplied to ct.gov.COG plans to submit data AE/SAE data consistent with the text in this field.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.